CLINICAL TRIAL: NCT05635253
Title: Influence of Polishing After Bleaching on Color Change and Enamel Morphology: Randomized Clinical Trial
Brief Title: Influence of Polishing After Bleaching on Color Change and Enamel Morphology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: UFPara-0014
Record Dates: First submitted 2022-11-13; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Tooth Discoloration; Morphologic Change; Tooth Sensitivity
MeSH Terms: conditions — Tooth Discoloration; Dentin Sensitivity | interventions — Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP GSEM (Other): In-office whitening treatment with 35% Hydrogen Peroxide
  Interventions: Other: Hydrogen Peroxide 35%
- GROUP GP (Experimental): In-office whitening treatment with 35% Hydrogen Peroxide + Polishing of whitened teeth
  Interventions: Other: Hydrogen Peroxide 35% + Polishing whitened teeth

INTERVENTIONS:
Other: Hydrogen Peroxide 35% — Group that received only bleaching treatment. Soft tissue protection was performed with a Top Dam light-curing gingival barrier (FGM, Santa Catarina, SC, Brazil). Application of whitening gel (Whitness HP 35%/FGM) on the buccal surface from premolar to premolar in the upper and lower arches. Three 45-minute sessions were held with an interval of seven days between them.
  Arms: GROUP GSEM
Other: Hydrogen Peroxide 35% + Polishing whitened teeth — Group that received only bleaching treatment followed by polishing. Soft tissue protection was performed with a Top Dam light-curing gingival barrier (FGM, Santa Catarina, SC, Brazil). Application of whitening gel (Whitness HP 35%/FGM) on the buccal surface from premolar to premolar in the upper and lower arches. Three 45-minute sessions were held with an interval of seven days between them. After bleaching, the vestibular surfaces were polished for 20s on each bleached tooth, with polishing paste and felt disc (Diamond Flex, FGM, Santa Catarina, SC, Brazil) in low rotation.
  Arms: GROUP GP

SUMMARY:
This trial evaluated the influence of polishing on enamel color change after in-office bleaching treatment. It also evaluated the influence of polishing on tooth morphology and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 30 years old of both sexes;
* With good oral hygiene;
* With no sensitivity to tactile and evaporative stimuli;
* Who have not undergone previous bleaching treatment, and with no caries lesions.

Exclusion Criteria:

* patients undergoing fixed orthodontic treatment;
* patients allergic to the bleaching product;
* drug users or pregnant women;
* patients with carious lesions, defective restorations and/or periodontal disease, patients with systemic diseases, pulpitis or patients using analgesics.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Influence of polishing on color after tooth whitening | 14 days
  Color evaluation was performed with the EasyshadeAdvanced spectrophotometer (Vita-Zahnfabrik, GE, Germany)

SECONDARY OUTCOMES:
Surface morphology of whitening enamel with and without polishing | 14 days
  The images were obtained using a electron microscope (Mira3 model) with type electron gun, mounted on supports of aluminum with 12mm of diameter, using tape double adhesive carbon face, and metallic with Au for 2'30'' which deposits about the sample a film thick average of 10 to 15nm. The images were generated by detecting secondary electrons, using a voltage acceleration of 5 kV and a working distance of around 15 mm.
Influence of polishing on sensitivity after tooth whitening | 14 days
  assessment of sensitivity during treatment using a visual analogue scale with values from 0 to 10, with higher values indicating a worse level of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Cecy Martins Silva, Belém, Pará, Brazil